CLINICAL TRIAL: NCT00722774
Title: Phase I Inpatient Study of the Safety and Immunogenicity of Live Influenza A Vaccine H2N2 (A/Ann Arbor/6/60 ca Recombinant), a Live Attenuated Virus Vaccine Candidate for Prevention of Influenza H2N2 Infection in the Event of a Pandemic
Brief Title: Safety and Immune Response to Recombinant Live-Attenuated Influenza H2N2 Virus Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Kawsar Talaat, MD, Johns Hopkins Bloomberg School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 247
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2008-11-10 (Estimated); Status verified 2008-07

CONDITIONS: Influenza; Virus Diseases
Keywords: Vaccine; Influenza
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Participants will receive 2 doses of vaccine 4 to 8 weeks (28-62 days) apart
  Interventions: Biological: H2N2 1960 AA ca recombinant vaccine

INTERVENTIONS:
Biological: H2N2 1960 AA ca recombinant vaccine — Approximately 0.2 ml of 10^7 TCID50 doses of vaccine administered intranasally

SUMMARY:
In the 20th century, influenza pandemics occurred in 1918, 1957, and 1968, and were associated with significant morbidity and mortality. It is estimated that, in the United States alone, the next influenza pandemic could cause approximately 200,000 deaths and 750,000 hospitalizations. Thus, the development of a vaccine against potential influenza strains has become a priority. The purpose of this study is to determine the safety and immune response to an H2N2 influenza vaccine candidate.

DETAILED DESCRIPTION:
H2N2 influenza viruses emerged in the 1950s replacing the then circulating H1N1 human influenza virus. The first cases occurred in China in 1956, and disease became widespread in 1956-1957, resulting in the "Asian Influenza" pandemic that was responsible for between 1 and 4 million deaths worldwide. H2N2 viruses have not circulated since 1968, when they were replaced by H3N2 influenza viruses and the resurgence of H1N1 viruses. For this reason, a large proportion of the population is now susceptible to infection with H2N2 influenza. If this subtype re-emerges, it could potentially cause the next pandemic. This vaccine, therefore, is an important priority in the development of vaccines against potential pandemic influenza strains.

This vaccine trial will be conducted in the Center for Immunization Research isolation unit in the Mason F. Lord Building at the Johns Hopkins Bayview Medical Center (Baltimore, MD). The study will be initiated between April 1st and December 20th, 2008, when wild-type influenza is unlikely to be circulating in the Baltimore area.

An individual's participation in the study will last approximately 90 days. All participants will receive two vaccinations approximately 4 - 8 weeks apart. After each vaccination, participants will remain in isolation at the study site for at least nine days or until rRT-PCR assays for influenza are negative for 2 consecutive days. A physical examination and nasal wash will occur each day during the isolation period. Blood collection will occur in isolation beginning on Day 7 until release. Follow-up outpatient visits are scheduled on Days 28 and 56 after the first vaccination and on Day 28 after the second vaccination. Follow-up visits will include serum collection, nasal wash, and interim medical history.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* Available for the duration of the trial
* If female, agree to use effective birth control methods for the duration of the study. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease. More information on this criterion can be found in the protocol.
* Behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, intereferes with the study
* Previous receipt of FluMist or any intranasal live attenuated influenza vaccine
* Previous enrollment in an H2N2 influenza vaccine trial or in any study of an avian influenza vaccine
* Seropositive to the H2N2 influenza A virus (serum HAI titer >1:8)
* Positive urine drug toxicology test indicating narcotic use and/or dependency as defined by the Drug Enforcement Agency
* Medical, occupational, or family problems as a result of alcohol or illicit drug use within the 12 months prior to study entry
* Any condition that, in the opinion of the investigator, would interfere with the study
* History of anaphylaxis
* Allergy to oseltamivir as determined by subject report
* Current diagnosis of asthma or reactive airway disease within 2 years prior to study entry
* History of Guillain-Barre Syndrome
* HIV-1-infected
* Hepatitis C-infected
* Positive hepatitis B virus surface antigen
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical preparations) or immunosuppressive drugs within 30 days prior to study entry
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to study entry
* History of a surgical splenectomy
* Receipt of blood or blood-derived products (including immunoglobulin) within 6 months prior to study entry
* Current smoker unwilling to stop smoking for the duration of the study. More information on this criterion can be found in the protocol.
* Travel to the Southern Hemisphere within 14 days prior to study entry
* Travel on a cruise ship within 14 days prior to study entry
* Direct contact with live poultry within the 14 days prior to the study or after study completion.
* Receipt of another investigational vaccine or drug within 30 days prior to study entry
* Allergy to eggs or egg products
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related reactogenicity events and other adverse events | Throughout study
Amount of vaccine virus shed by each participant | Throughout study
Amount of serum and nasal wash antibody induced by the vaccine | Throughout study

SECONDARY OUTCOMES:
Number of participants infected with the H2N2 1960 AA ca recombinant vaccine | Throughout study
Phenotypic stability of vaccine virus shed | Throughout study
Determine whether immunogenicity is enhanced by a second dose of vaccine, and whether the first dose of vaccine restricts replication of the second dose | Throughout study
T-cell mediated and innate immune responses against the H2N2 1960 AA ca recombinant vaccine | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bayview Medical Center, CIR Unit at the Mason F Lord Building, Baltimore, Maryland, United States

REFERENCES:
- [Background] Eichelberger M, Golding H, Hess M, Weir J, Subbarao K, Luke CJ, Friede M, Wood D. FDA/NIH/WHO public workshop on immune correlates of protection against influenza A viruses in support of pandemic vaccine development, Bethesda, Maryland, US, December 10-11, 2007. Vaccine. 2008 Aug 12;26(34):4299-303. doi: 10.1016/j.vaccine.2008.06.012. Epub 2008 Jun 26. PMID 18582523
- [Background] Hampson AW. Vaccines for pandemic influenza. The history of our current vaccines, their limitations and the requirements to deal with a pandemic threat. Ann Acad Med Singap. 2008 Jun;37(6):510-7. PMID 18618064
- [Background] Wright PF. Vaccine preparedness--are we ready for the next influenza pandemic? N Engl J Med. 2008 Jun 12;358(24):2540-3. doi: 10.1056/NEJMp0803650. No abstract available. PMID 18550873